CLINICAL TRIAL: NCT01569295
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Idelalisib (GS-1101) in Combination With Bendamustine and Rituximab for Previously Treated Chronic Lymphocytic Leukemia
Brief Title: Study Evaluating the Efficacy and Safety of Idelalisib in Combination With Bendamustine and Rituximab for Previously Treated Chronic Lymphocytic Leukemia (CLL) (Tugela )
Acronym: Tugela
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-312-0115; 2011-006292-20 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-04-03 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Zydelig; CLL; CAL-101; GS 1101; GS-1101; PI3K; Rituxan; Rituximab; Bendamustine; Leukemia; idelalisib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — idelalisib; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Idelalisib+bendamustine+rituximab (Experimental): Participants will receive idelalisib plus bendamustine and rituximab
  Interventions: Drug: Idelalisib; Drug: Rituximab; Drug: Bendamustine
- Placebo to match idelalisib+bendamustine+rituximab (Placebo Comparator): Participants will receive placebo to match idelalisib plus bendamustine and rituximab
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Placebo to match idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib 150 mg administered orally twice daily
  Other Names: GS-1101; CAL-101; Zydelig®
  Arms: Idelalisib+bendamustine+rituximab
Drug: Rituximab — Rituximab 375 mg/m^2 on Day 1, then 500 mg/m^2 every 28 days administered intravenously for a maximum of 6 infusions
  Other Names: Rituxan®; MabThera
Drug: Bendamustine — Bendamustine 70 mg/mg^2/day on 2 consecutive days every 28 days administered intravenously for a maximum of 12 infusions
  Other Names: Ribomustin; Treanda®
Drug: Placebo to match idelalisib — Placebo to match idelalisib administered orally twice daily
  Arms: Placebo to match idelalisib+bendamustine+rituximab

SUMMARY:
The primary objective of this study is to evaluate the effect of the addition of idelalisib (formerly GS-1101) to bendamustine + rituximab (BR) on progression-free survival (PFS) in participants with previously treated chronic lymphocytic leukemia (CLL)

ELIGIBILITY:
Key Inclusion Criteria:

* Previously treated recurrent CLL
* Measurable lymphadenopathy
* Requires therapy for CLL
* Has experienced CLL progression < 36 months since the completion of the last prior therapy

Key Exclusion Criteria:

* Recent history of a major non-CLL malignancy
* Evidence of an ongoing infection
* CLL refractory to bendamustine
* Concurrent participation in another therapeutic clinical trial

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (106):
- United States (23):
  - Clearview Cancer Institute, Huntsville, Alabama
  - UCLA Medical Center, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Summit Medical Group, P.A., Morristown, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Texas Oncology, Austin, Texas
  - Texas Oncology PA, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Cancer Care Northwest, US Oncology, Spokane, Washington
  - Virginia Cancer Specialists, PC, Vancouver, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - St Vincent's Hospital - Sydney, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre - Clayton Campus, Clayton, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (3):
  - Ziekenhuisnetwerk Antwerpen - AZ Stuivenberg, Antwerp
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Cancer Care Manitoba, Winnipeg, Manitoba, Canada
- Croatia (3):
  - Clinical Hospital "Dubrava", Zagreb
  - Klinichki Bolnicki Centar-Zagreb, Zagreb
  - University Hospital Merkur, Zagreb
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava
- France (9):
  - Hopital Henri Mondor, Créteil
  - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - CHRU Lille-Hôpital Claude Huriez, Lille
  - Centre Léon Bérard - Centre régional de lutte contre le cancer Rhône-Alpes, Lyon
  - Centre Hospitalier de Mulhouse, Mulhouse
  - CHU Hôtel-Dieu-Service Hématologie, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Purpan, Toulouse
  - Hôpitaux de Brabois, Vandoeuvre-lés-Nancy
- Greece (2):
  - G. Genimatas Hospital, Athens
  - University General Hospital of Patras, Pátrai
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Debrecen
  - Tallian Gyula utca 20-32, Kaposvár
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Mater Misericordiae Hospital, Dublin, Ireland
- Italy (4):
  - Spedali Civili di Brescia, Brescia
  - Ospedale Oncologico Regionale A. Businco, Cagliari
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria San Giovanni Battista-Molinette, Torino
- Poland (7):
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Malopolskie Centrum Medyczne, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Wojewodzki Szpital w Opolu, Opole
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Warsaw
- Portugal (2):
  - Hospital Santa Maria, Lisbon
  - "Instituto Portugues de Oncologia do Porto Francisco Gentil (IPOPFG, EPE), Porto
- Romania (4):
  - Emergency County Clinical Hospital Brasov, Brasov
  - "Colentina" Clinical Hospital, Bucharest
  - "Fundeni" Clinical Institute, Bucharest
  - Regional Oncology Institute Iasi, Iași
- Russia (7):
  - Russian Oncology Research Center (N.N. Blokhin), Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. N.A. Semashko, Nizhny Novgorod
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Ryazan Regional Clinical Hospital, Ryazan
  - Research Institute of Hematology and Blood Transfusion, Saint Petersburg
  - Saratov State Medical University, Saratov
  - State Budgetary Healthcare Institution Volgograd Regional Clinical Oncology Dispensary #1, Volgograd
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital 12 de Octubre, Madrid, Madrid, Communidad de
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid, Communidad de
  - Hospital Universitario de La Princesa, Madrid
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty Gazi Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Ondokuz Mayis University Faculty of Medicine, Samsun
- United Kingdom (15):
  - Birmingham Heartlands Hospital, Birmingham
  - Kent and Canterbury Hospital, Canterbury
  - University Hospital of Wales, Cardiff
  - Dorset County Hospital, Dorchester
  - St. James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - St Bartholomews Hospital, London
  - King's College Hospital, London
  - Hammersmith Hospital, London
  - University College London, London
  - Christie Hospital, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Churchill Hospital, Oxford
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Background] Zelenetz AD, Robak T, et al. Idelalisib Plus Bendamustine and Rituximab (BR) Is Superior to BR Alone in Patients with Relapsed/Refractory Chronic Lymphocytic Leukemia: Results of a Phase 3 Randomized Double-Blind Placebo-Controlled Study. American Society ofHematology (ASH) 57th Annual Meeting & Exposition; 5-8 December 2015; Orlando, FL.
- [Background] Barrientos JC, Brown JR, et al. Results of a Randomized Double-Blind Placebo-Controlled Phase 3 study Evaluating Idelalisib in Combination with Bendamustine and Rituximab in Patients with Relapsed/Refractory CLL and Adverse Prognostic Features. American Society of Clinical Oncology (ASCO) 2016 Annual Meeting; 3-7 June 2016; Chicago, IL.
- [Background] Hillmen, P, Ferra C, et al. Idelalisib in Combination with Bendamustine and Rituximab Improves Overall Survival in Patients with Relapsed/Refractory CLL: Interim Results of a Phase 3 Randomized Double-Blind Placebo-Controlled Study. European Hematology Association (EHA) 21st Annual Meeting; 9-12 June 2016; Copenhagen, Denmark.
- [Background] Zelenetz AD, Brown JR et al. Updated Analysis of Overall Survival in Randomized Phase III Study of Idelalisib in Combination with Bendamustine and Rituximab in Patients with Relapsed/Refractory CLL. American Society of Hematology (ASH) 58th Annual Meeting & Exposition; 3-6 December 2016; San Diego, CA
- [Background] Zelenetz AD, Barrientos JC, Brown JR, Coiffier B, Delgado J, Egyed M, Ghia P, Illes A, Jurczak W, Marlton P, Montillo M, Morschhauser F, Pristupa AS, Robak T, Sharman JP, Simpson D, Smolej L, Tausch E, Adewoye AH, Dreiling LK, Kim Y, Stilgenbauer S, Hillmen P. Idelalisib or placebo in combination with bendamustine and rituximab in patients with relapsed or refractory chronic lymphocytic leukaemia: interim results from a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2017 Mar;18(3):297-311. doi: 10.1016/S1470-2045(16)30671-4. Epub 2017 Jan 28. PMID 28139405
- [Derived] Montillo M, Illes A, Robak T, Pristupa AS, Wach M, Egyed M, Delgado J, Jurczak W, Morschhauser F, Schuh A, Eradat H, Shreay S, Barrientos JC, Zelenetz AD. Idelalisib addition has neutral to beneficial effects on quality of life in bendamustine/rituximab-treated patients: results of a phase 3, randomized, controlled trial. Health Qual Life Outcomes. 2019 Nov 15;17(1):173. doi: 10.1186/s12955-019-1232-8. PMID 31729982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 110 sites in Australia, New Zealand, Europe, Asia and North America. The first participant was screened on 15 June 2012. The last study visit occurred on 10 June 2019.
Pre-assignment Details: 540 participants were screened.
Groups:
- Idelalisib + Bendamustine + Rituximab: Idelalisib 150 mg tablet administered orally twice daily (until the earliest of participant withdrawal from study, definitive progression of chronic lymphocytic leukemia (CLL), intolerable toxicity, pregnancy, substantial noncompliance with study procedures, or study discontinuation) + rituximab 375 mg/m^2 on Day 1, then 500 mg/m^2 every 28 days administered intravenously for a total of 6 infusions + bendamustine 70 mg/mg^2/infusion on days 1 and 2 of each 28 day cycle, administered intravenously for a total of 6 cycles (12 infusions).
- Placebo + Bendamustine + Rituximab: Placebo to match idelalisib administered orally twice daily + rituximab 375 mg/m^2 on Day 1, then 500 mg/ m^2 every 28 days administered intravenously for a total of 6 infusions + bendamustine 70 mg/m^2/infusion on days 1 and 2 of each 28 day cycle administered intravenously for a total of 6 cycles (12 infusions).
Period: Overall Study
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Started | 207 | 209
Long-Term Follow-up | 109 | 161
Completed | 0 | 0
Not Completed | 207 | 209
Not completed — Progressive Disease | 75 | 139
Not completed — Adverse Event | 39 | 14
Not completed — Withdrawal by Subject | 25 | 12
Not completed — Death | 19 | 15
Not completed — Physician Decision | 13 | 18
Not completed — Study Terminated by Sponsor | 24 | 2
Not completed — Other Reason not Specified | 3 | 5
Not completed — Non-Compliance with Study Drug | 6 | 1
Not completed — Other Anticancer/Experimental Therapy | 2 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) Analysis Set included all participants randomized in the study regardless of whether study drug was administered and with treatment group designated according to initial randomization.
Groups:
- Idelalisib + Bendamustine + Rituximab: Idelalisib 150 mg tablet administered orally twice daily (until the earliest of participant withdrawal from study, definitive progression of CLL, intolerable toxicity, pregnancy, substantial noncompliance with study procedures, or study discontinuation) + rituximab 375 mg/m^2 on Day 1, then 500 mg/m^2 every 28 days administered intravenously for a total of 6 infusions + bendamustine 70 mg/mg^2/infusion on days 1 and 2 of each 28 day cycle, administered intravenously for a total of 6 cycles (12 infusions).
- Total: Total of all reporting groups
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab | Total
Number analyzed (Participants) | 207 | 209 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9.2) | 63 (9.8) | 62 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 53 | 100
  Male | 160 | 156 | 316
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 187 | 190 | 377
  Race: Black or African American | 6 | 4 | 10
  Race: Asian | 2 | 1 | 3
  Race: Other | 2 | 2 | 4
  Race: Not Permitted | 10 | 12 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 4 | 5 | 9
  Ethnicity: Not Hispanic or Latino | 191 | 188 | 379
  Ethnicity: Not Permitted | 12 | 15 | 27
  Ethnicity: Missing | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 5 | 6 | 11
  Hungary | 24 | 20 | 44
  United States | 37 | 33 | 70
  Czechia | 9 | 5 | 14
  United Kingdom | 27 | 29 | 56
  Portugal | 1 | 4 | 5
  Russia | 22 | 14 | 36
  Spain | 14 | 18 | 32
  Greece | 1 | 1 | 2
  Canada | 0 | 3 | 3
  Turkey | 6 | 6 | 12
  Belgium | 3 | 7 | 10
  Ireland | 1 | 1 | 2
  Poland | 17 | 22 | 39
  Italy | 10 | 7 | 17
  Australia | 8 | 8 | 16
  France | 13 | 14 | 27
  Croatia | 5 | 9 | 14
  New Zealand | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the interval from randomization to the earlier of the first documentation of definitive disease progression or death from any cause. PFS (months) = (minimum (date of disease progression, date of death) - date of randomization + 1)/30.4375.
Time Frame: Up to 84 months
Population: The intent-to-treat (ITT) Analysis Set included all participants randomised in the study regardless of whether study drug was administered and with treatment group designated according to initial randomisation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 207 | 209
months | 21.8 [16.5 to 27.8] | 11.1 [8.9 to 11.1]
Statistical Analysis 1: Comparison: Idelalisib + Bendamustine + Rituximab vs Placebo + Bendamustine + Rituximab; Test type: Superiority; p < 0.0001, Stratified log-rank test; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.27 to 0.45] — Hazard Ratio is estimated using Cox proportional hazard model, adjusted for randomization stratification factors

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was the percentage of participants who achieved a complete response (CR), CR with incomplete marrow recovery (CRi,) or partial response (PR) and maintained the response for at least 12 weeks. CR was defined as no lymphadenopathy, hepatomegaly, splenomegaly; normal complete blood count; confirmed by bone marrow aspirate & biopsy.
  PR was defined as >1 of the following criteria: a 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver size, spleen size; plus ≥ 1 of the following: ≥ 1500/μL absolute neutrophil count, > 100000/μL platelets, > 11.0 g/dL hemoglobin or 50% improvement for either of these parameters without transfusions or growth factors. CRi was defined as all criteria for CR met but with persistent anemia, thrombocytopenia, neutropenia or a hypocellular bone marrow.
Time Frame: Up to 84 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 207 | 209
percentage of participants | 70.0 [63.3 to 76.2] | 45.5 [38.6 to 52.5]
Statistical Analysis 1: Comparison: Idelalisib + Bendamustine + Rituximab vs Placebo + Bendamustine + Rituximab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Odds ratio,p-value and 95% Confidence Interval(CI) were calculated from Cochran-Mantel-Haenszel(CMH) Chi-square test stratified by stratification factor in EDC(del17p/TP53,immunoglobulin heavy chain variable region(IgHV) mutation and disease status); Odds Ratio (OR) = 3.02, 95% CI 2-sided [1.98 to 4.62]

3. Secondary Outcome: Lymph Node Response Rate
Description: Lymph node response rate was defined as the percentage of participants who achieved a ≥ 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters (SPD) of index lesions.
Time Frame: Up to 84 months
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 192 | 197
percentage of particpants | 96.9 [93.3 to 98.8] | 60.9 [53.7 to 67.8]
Statistical Analysis 1: Comparison: Idelalisib + Bendamustine + Rituximab vs Placebo + Bendamustine + Rituximab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Odds ratio, p-value and 95% CI were calculated from the CMH Chi-square test stratified by stratification factors in EDC (del17p/TP53, IgHV mutation and disease status); Odds Ratio (OR) = 28.81, 95% CI 2-sided [10.50 to 79.02]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the interval from randomization to death from any cause. Overall survival (months) = (date of death - date of randomization + 1)/30.4375.
Time Frame: Up to 84 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 207 | 209
months | 56.2 [40.1 to NA] — Upper CI was not reached due to the low number of deaths by the time of study closure. | 42.6 [35.3 to 54.8]
Statistical Analysis 1: Comparison: Idelalisib + Bendamustine + Rituximab vs Placebo + Bendamustine + Rituximab; Test type: Superiority; p = 0.098, Stratified log-rank test; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.59 to 1.03]

5. Secondary Outcome: Complete Response Rate
Description: Complete response (CR) rate was defined as the percentage of participants who achieved a CR.
Time Frame: Up to 84 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
Number analyzed (Participants) | 207 | 209
percentage of participants | 4.3 [2.0 to 8.1] | 0.5 [0 to 2.6]
Statistical Analysis 1: Comparison: Idelalisib + Bendamustine + Rituximab vs Placebo + Bendamustine + Rituximab; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel — Odds ratio, 95% CI and p-value are calculated from the CMH Chi-square test stratified by stratification factors in EDC (del17p/TP53, IgHV mutation and disease status); Odds Ratio (OR) = 9.55, 95% CI 2-sided [1.19 to 76.81]

ADVERSE EVENTS:
Time Frame: First dose up to the last dose date plus 30 days (Up to approximately 67.7 months)
Description: The Safety Analysis Set included all participants who received >=1 dose of study treatment, with treatment group assignments designated according to the actual treatment received.
Arm/Group | Idelalisib + Bendamustine + Rituximab | Placebo + Bendamustine + Rituximab
All-Cause Mortality (participants affected / at risk) | 89/207 | 106/209
Serious Adverse Events (participants affected / at risk) | 152/207 | 94/209
Other Adverse Events (participants affected / at risk) | 199/207 | 196/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Bendamustine + Rituximab (N=207) | Placebo + Bendamustine + Rituximab (N=209)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 8 | 5
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 45 | 10
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 9 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Rhegmatogenous retinal detachment (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Ascites (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 5 | 1
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Pyrexia (General disorders) | 25 | 11
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Biliary fistula (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Aspergillus infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 5
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 4 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 1
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Cytomegalovirus enteritis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 3 | 1
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Ecthyma (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 2 | 0
Eye infection toxoplasmal (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis cryptosporidial (Infections and infestations) | 1 | 0
H1n1 influenza (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 4 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 3 | 1
Lower respiratory tract infection (Infections and infestations) | 7 | 5
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 3
Meningitis aseptic (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Meningitis enteroviral (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 6
Ophthalmic herpes zoster (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 0
Oropharyngitis fungal (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 2
Perineal infection (Infections and infestations) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 38 | 16
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 1
Pneumonia pseudomonal (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 5 | 5
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 11 | 4
Septic shock (Infections and infestations) | 5 | 1
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 3
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Bk polyomavirus test positive (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Streptococcus test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Reiter's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 1 | 0
Perineal necrosis (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Bendamustine + Rituximab (N=207) | Placebo + Bendamustine + Rituximab (N=209)
Anaemia (Blood and lymphatic system disorders) | 54 | 48
Leukopenia (Blood and lymphatic system disorders) | 17 | 10
Neutropenia (Blood and lymphatic system disorders) | 129 | 113
Thrombocytopenia (Blood and lymphatic system disorders) | 41 | 46
Abdominal pain (Gastrointestinal disorders) | 21 | 13
Constipation (Gastrointestinal disorders) | 32 | 35
Diarrhoea (Gastrointestinal disorders) | 89 | 47
Dyspepsia (Gastrointestinal disorders) | 15 | 8
Nausea (Gastrointestinal disorders) | 60 | 72
Vomiting (Gastrointestinal disorders) | 35 | 31
Asthenia (General disorders) | 24 | 20
Chills (General disorders) | 22 | 13
Fatigue (General disorders) | 45 | 52
Oedema peripheral (General disorders) | 17 | 18
Pyrexia (General disorders) | 78 | 55
Hypogammaglobulinaemia (Immune system disorders) | 12 | 10
Bronchitis (Infections and infestations) | 20 | 8
Herpes zoster (Infections and infestations) | 11 | 6
Lower respiratory tract infection (Infections and infestations) | 13 | 10
Nasopharyngitis (Infections and infestations) | 16 | 11
Pneumonia (Infections and infestations) | 25 | 13
Respiratory tract infection (Infections and infestations) | 7 | 11
Sinusitis (Infections and infestations) | 19 | 13
Upper respiratory tract infection (Infections and infestations) | 37 | 21
Infusion related reaction (Injury, poisoning and procedural complications) | 29 | 45
Alanine aminotransferase increased (Investigations) | 32 | 2
Aspartate aminotransferase increased (Investigations) | 19 | 2
Weight decreased (Investigations) | 25 | 12
Decreased appetite (Metabolism and nutrition disorders) | 24 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 15
Headache (Nervous system disorders) | 20 | 21
Anxiety (Psychiatric disorders) | 6 | 12
Insomnia (Psychiatric disorders) | 19 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 26
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 | 12
Night sweats (Skin and subcutaneous tissue disorders) | 18 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 12
Rash (Skin and subcutaneous tissue disorders) | 36 | 28
Hypertension (Vascular disorders) | 13 | 5
Hypotension (Vascular disorders) | 14 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT01569295/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT01569295/SAP_001.pdf